CLINICAL TRIAL: NCT05476796
Title: Randomised Phase II Study Evaluating Trifluridine/Tipiracil Plus Oxaliplatin ± Nivolumab Versus FOLFOX ± Nivolumab in Patients With HER2 Negative Locally Advanced, Recurrent or Metastatic Gastric, Oesophageal or Oesogastric Junction Adenocarcinoma
Brief Title: Oxaliplatin ± Nivolumab in Combination With Trifluridine/Tipiracil or 5-fluorouracile in Frail Patients With Advanced, Recurrent or Metastatic Gastric, Oesophageal or Gastroesophageal Junction Cancer
Acronym: LOGICAN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Servier (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-GIG-2203; 2022-000273-81 (EudraCT Number); 2024-512999-35-00 (EU CTIS Number)
Record Dates: First submitted 2022-07-26; First posted 2022-07-27 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Gastric Adenocarcinoma; Esophagus Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
Keywords: Metastatic; Recurrent; Locally advanced; Trifluridine/Tipiracil; Gastrointestinal; Adenocarcinoma; FOLFOX; Oxaliplatin; Gastric Adenocarcinoma; Esophagus Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Gastric; Esophagus; Gastroesophageal Junction
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Neoplasm Metastasis; Recurrence; Adenocarcinoma | interventions — trifluridine tipiracil drug combination; Oxaliplatin; Folfox protocol; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trifluridine/Tipiracil + Oxaliplatin ± nivolumab (Experimental): Trifluridine/Tipiracil will be administered with a 14-day schedule (35 mg/m² twice-daily [BID] for 5 days followed by 9 days of recovery) until disease progression or intolerable toxicity.
  Oxaliplatin will be administered intravenously on day 1 of each treatment cycle (infusion duration: 2 hours), every 2 weeks. The first cycle will be administered at level -1 (70 mg/m²) and then increased to 85 mg/m² (if feasible) from the cycle 2 to 8 or until disease progression, whatever occurs first. In case of limiting-oxaliplatin neuropathy and in all cases after 8 cycles, oxaliplatin will be stopped and Trifluridine/Tipiracil will be continued alone until disease progression or intolerable toxicity.
  ± nivolumab 240 mg (infusion duration 30 minutes, every 2 weeks) until disease progression or intolerable toxicity for a maximum of 2 years.
  Interventions: Drug: Trifluridine/Tipiracil; Drug: Oxaliplatin; Drug: Nivolumab
- FOLFOX ± nivolumab (Active Comparator): Folinic Acid 400 mg/m² (or 200 mg/m² if L-folinic acid) + oxaliplatin 85 mg/m² (infusion duration: 2 hours) followed by 5-FU bolus 400 mg/m² and then 5-FU 2400 mg/m² as a 46-hour continuous infusion. Treatment repeated every 14 days. In case of limiting-oxaliplatin neuropathy and in all cases after 8 cycles, oxaliplatin will be stopped and 5-FU (simplified LV5FU2 regimen) or capecitabine (1000 mg/m² BID during 2 weeks every 3 weeks) will be continued alone until disease progression or intolerable toxicity.
  ± nivolumab 240 mg (infusion duration 30 minutes, every 2 weeks) until disease progression or intolerable toxicity for a maximum of 2 years.
  Interventions: Drug: FOLFOX regimen; Drug: Nivolumab

INTERVENTIONS:
Drug: Trifluridine/Tipiracil — Trifluridine/Tipiracil will be administered with a 14-day schedule (35 mg/m² BID for 5 days followed by 9 days of recovery) until disease progression or intolerable toxicity.
  Other Names: Lonsurf
  Arms: Trifluridine/Tipiracil + Oxaliplatin ± nivolumab
Drug: Oxaliplatin — Oxaliplatin will be administered intravenously on day 1 of each treatment cycle (infusion duration: 2 hours), every 2 weeks. The first cycle will be administered at level -1 (70 mg/m²) and then increased to 85 mg/m² (if feasible) from the cycle 2 to 8 or until disease progression, whatever occurs first. In case of limiting-oxaliplatin neuropathy and in all cases after 8 cycles, oxaliplatin will be stopped and Trifluridine/Tipiracil will be continued alone until disease progression or intolerable toxicity.
  Arms: Trifluridine/Tipiracil + Oxaliplatin ± nivolumab
Drug: FOLFOX regimen — Folinic Acid 400 mg/m² (or 200 mg/m² if L-folinic acid) + oxaliplatin 85 mg/m² (infusion duration: 2 hours) followed by 5-FU bolus 400 mg/m² and then 5-FU 2400 mg/m² as a 46-hour continuous infusion. Treatment repeated every 14 days. In case of limiting-oxaliplatin neuropathy and in all cases after 8 cycles, oxaliplatin will be stopped and 5-FU (simplified LV5FU2 regimen) or capecitabine (1000 mg/m² BID during 2 weeks every 3 weeks) will be continued alone until disease progression or intolerable toxicity.
  Arms: FOLFOX ± nivolumab
Drug: Nivolumab — Nivolumab 240 mg (infusion duration 30 minutes, every 2 weeks) until disease progression or intolerable toxicity for a maximum of 2 years
  Other Names: OPDIVO

SUMMARY:
Oxaliplatin ± nivolumab in combination with trifluridine/tipiracil or 5-fluorouracile (5-FU) in frail patients with advanced, recurrent or metastatic gastric, oesophageal or gastroesophageal junction cancer.

DETAILED DESCRIPTION:
Randomised Phase II Study Evaluating Trifluridine/Tipiracil Plus Oxaliplatin ± Nivolumab Versus FOLFOX ± Nivolumab in Patients With HER2 Negative Locally Advanced, Recurrent or Metastatic Gastric, Oesophageal or Oesogastric Junction Adenocarcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed locally advanced, recurrent or metastatic non resectable adenocarcinoma of the stomach, oesophagus or gastroesophageal junction (GEJ) ineligible to curative treatment.
2. No dysphagia or difficulty in swallowing.
3. No overexpression/amplification of HER2 (IHC 0 or 1+; if IHC is 2+, HIS must be negative). Known combined positive scor (CPS) PD-L1 score (result in % with the name of the method used). The microsatellite and mismatch repair (MMR) status of patient's tumour (MSI/MSS and pMMR/dMMR) must also be known at the time of screening (IHC and PCR tests have to be done).
4. At least one evaluable lesion according to RECIST v1.1 outside any previously irradiated area.
5. No prior palliative chemotherapy.
6. Age ≥18 years old.
7. Patient eligible for FOLFOX chemotherapy
8. Adequate organs function:

   * Absolute neutrophils count ≥1.5x10⁹/L
   * Platelets count ≥100x10⁹/L
   * Haemoglobin ≥9 g/L
   * Serum bilirubin levels <2 times upper limit of normal (ULN), up to 2.5 times ULN in case of hepatic metastasis (biliary drainage allowed)
   * Transaminases <5 times ULN
   * Creatinine clearance >40 mL/min
9. No Dihydropyrimidine dehydrogenase (DPD) deficiency (uracilemia <16 ng/ml)
10. Women of childbearing potential must have a negative serum or urine pregnancy test done within 14 days before the first study treatment.
11. Patients must agree to use adequate contraception methods for the duration of study treatment and within 6 months after completing treatment.
12. Patients must be affiliated to a Social Security System (or equivalent).
13. Patient must have signed and dated a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent.
14. Availability of archived tumour material for ancillary studies

Exclusion Criteria:

1. Patient with a performance status ECOG PS >2.
2. Other current or previous malignancy within the past 3 years (with the exception of squamous cell carcinoma of the skin treated by surgery).
3. Adjuvant chemotherapy or radio-chemotherapy completed for less than 6 months.
4. Peripheral neuropathy of NCI-CTCAE grade ≥2 at baseline.
5. Patients with known allergy or severe hypersensitivity to any of the trial drugs or any of the trial drug excipients.
6. Patients unwilling or unable to comply with trial obligations for geographic, social, or physical reasons, or who are unable to understand the purpose and procedures of the trial.
7. Previous treatment with trifluridine/tipiracil.
8. Known Human Immunodeficiency Virus (HIV) infection.
9. Active Hepatitis B virus (HBV, defined as having a positive hepatitis B surface antigen [HBsAg] test prior to inclusion) or hepatitis C virus (HCV).
10. Interstitial lung disease.
11. Prior pneumonitis requiring systemic corticosteroid therapy.
12. Active infections.
13. Pregnant or breastfeeding woman.
14. Participation in another therapeutic trial within the 30 days prior to randomisation.
15. Persons deprived of their liberty or under protective custody or guardianship.
16. Clinically relevant coronary artery disease or history of myocardial infarction in the last 12 months, or high risk of uncontrolled arrhythmia (for men: QTc ≥450 msec, for women: QTc ≥470 msec)
17. Active systemic autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enrol.
18. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first study drug administration. Inhaled or topical steroids are permitted in the absence of active autoimmune disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Progression free-survival | From randomization to disease progression or death up to 5 years
  The progression-free survival (PFS) is the length of time during and after the treatment of a disease that a patient lives with the disease but it does not get worse.

SECONDARY OUTCOMES:
Objective response rate | 5 years
  Objective response rate (ORR) is defined as the percentage of patients with a best response during treatment being either Complete Response (CR) or Partial Response (PR).
Overall survival | From randomization to death from any cause, up to 5 years
  The overall survival (OS) is the length of time from randomization that patients enrolled in the study are still alive.
Incidence of Treatment Adverse Events | Throughout study completion, up to 5 years
  The tolerance and safety will be evaluated by toxicity (acute [<1 months after the end of the trial treatment] and late [≥1 month after the end of the trial treatment), assessed using the Common terminology criteria for adverse events version 5.0 (CTCAE v5.0). CTCAE is widely accepted in the community of oncology research as the leading rating scale for adverse events. This scale, divided into 5 grades (1 = "mild", 2 = "moderate", 3 = "severe", 4 = "life-threatening", and 5 = "death") determined by the investigator, will make it possible to assess the severity of the disorders.
Time to patient performance status deterioration >2 | From randomization to PS deterioration >2, up to 5 years
  Time to performance status (PS) deterioration >2 is defined as the time between patient randomisation and the first date when PS>2.
  The Eastern Cooperative Oncology Group (ECOG) PS, a simple measure of functional status, determines ability of patient to tolerate therapies. It has scores ranging from 0 to 5 (0 = "fully active", 1 = "completely ambulatory", 2 = "<50% in bed during the day", 3 = ">50% in bed, but not bedbound", 4 = "bedbound", and 5 = "death").
Quality of life questionnaire - Core 30 (QLQ-C30) | From baseline until disease progression, up to 1 year
  Developed by the EORTC, this self-reported questionnaire assesses the health-related quality of life of cancer patients in clinical trials.
  The questionnaire includes five functional scales (physical, everyday activity, cognitive, emotional, and social), three symptom scales (fatigue, pain, nausea and vomiting), a health/quality of life overall scale, and a number of additional elements assessing common symptoms (including dyspnea, loss of appetite, insomnia, constipation, and diarrhea), as well as, the perceived financial impact of the disease.
  All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.

CONTACTS AND LOCATIONS:
Overall Officials: Christelle DE LA FOUCHARDIERE, Principal Investigator — Institut Paoli-Calmettes
Locations (29):
- France (29):
  - Clinique de l'Europe, Amiens
  - Hopital Privé Arras Les Bonnettes, Arras
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier de Beauvais, Beauvais
  - CHU Besançon - Hôpital Jean Minjoz, Besançon
  - CHU Morvan, Brest
  - Clinique Pasteur Lanroze, Brest
  - CH Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - CHU d'Estaing, Clermont-Ferrand
  - Institut Andrée Dutreix - Clinique de Flandre, Coudekerque-Branche
  - Centre Georges François Leclerc, Dijon
  - Hôpital Nord-Ouest Villefranche-sur-Saône, Gleizé
  - Centre Léon Bérard, Lyon
  - Hôpital Saint Joseph, Marseille
  - Institut Paoli Calmettes, Marseille
  - Hôpital Nord Franche Comté, Montbéliard
  - Centre Antoine Lacassagne, Nice
  - Hôpital Saint Louis, Paris
  - Hopital Europeen Georges Pompidou, Paris
  - GH Diaconesses - Crois St Simon, Paris
  - Institut Mutualiste Montsouris, Paris
  - CHU de Poitiers, Poitiers
  - CHU - Hôpital Robert Debré, Reims
  - Institut Jean Godinot, Reims
  - CHU Rouen - Charles Nicolle, Rouen
  - ICO - Site René Gauducheau, Saint-Herblain
  - Institut de cancérologie Strasbourg Europe, Strasbourg
  - CHU Nancy - Hôpital Brabois, Vandœuvre-lès-Nancy

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- [Derived] Botsen D, Chabaud S, Perrier H, Ammarguellat H, Jestin-Le-Tallec V, Olesinski J, Toullec C, Aparicio T, Ben Abdelghani M, Borg C, Bouche O, Coutzac C, Devaud H, Di Fiore F, Dubreuil O, Evesque L, Huguenin B, Muller M, Poureau PG, Oularue E, Tougeron D, Zaanan A, Ammari S, De Sousa Carvalho N, Decazes P, De La Fouchardiere C. Trifluridine/tipiracil + oxaliplatin +/- nivolumab vs FOLFOX +/- nivolumab in HER2 negative advanced oesogastric adenocarcinoma: The PRODIGE73-UCGI40-LOGICAN trial. Dig Liver Dis. 2024 Aug;56(8):1281-1287. doi: 10.1016/j.dld.2024.04.032. Epub 2024 May 17. PMID 38762353